CLINICAL TRIAL: NCT05816902
Title: Development and Validation of an Artificial Intelligence Prediction Model and a Survival Risk Stratification for Lung Metastasis in Colorectal Cancer From Highly Imbalanced Data
Brief Title: AI Prediction Model and Risk Stratification for Lung Metastasis in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Xishan Wang, the Cancer Hospital Chinese Academy of Medical Sciences and Peking Union Medical College, Peking Union Medical College
Other Study IDs: PekingUMC02
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer; Lung Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- validation set 1: The validation set 1 was comprised of patients with CRC diagnosed and treated between January 1, 2016, and December 31, 2020, at the Cancer Hospital Chinese Academy of Medical Sciences and Peking Union Medical College.
  Interventions: Other: The location of the patient's treatment
- validation set 2: The validation set 2 was comprised of patients with CRC diagnosed and treated between January 1, 2016, and December 31, 2020, at the Second Affiliated Hospital of Harbin Medical University.
  Interventions: Other: The location of the patient's treatment

INTERVENTIONS:
Other: The location of the patient's treatment — The location of the patient's treatment

SUMMARY:
Background:

To assist clinicians with diagnosis and optimal treatment decision-making, we attempted to develop and validate an artificial intelligence prediction model for lung metastasis (LM) in colorectal cancer (CRC) patients.

Method:

The clinicopathological characteristics of 46037 CRC patients from the Surveillance, Epidemiology, and End Results (SEER) database and 2779 CRC patients from a multi-center external validation set were collected retrospectively. After feature selection by univariate and multivariate analyses, six machine learning (ML) models, including logistic regression, K-nearest neighbor, support vector machine, decision tree, random forest, and balanced random forest (BRF), were developed and validated for the LM prediction. The optimization model with best performance was compared to the clinical predictor. In addition, stratified LM patients by risk score were utilized for survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with pathologic confirmation of a primary CRC diagnosis

Exclusion Criteria:

* (1) patients with multiple primary cancers or other malignancies; (2) patients identified via autopsy or death certificate; and (3) patients with uncertain clinical data values

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with pathologic confirmation of a primary CRC diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 2779 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
lung metastasis | through study completion, an average of 3 month
  diagnosed with lung metastasis